CLINICAL TRIAL: NCT00025103
Title: Protocol For The Treatment Of Relapsed And Refractory Wilms Tumour And Clear Cell Sarcoma Of The Kidney (CCSK)
Brief Title: Chemotherapy Followed by Surgery and Radiation Therapy With or Without Stem Cell Transplant in Treating Patients With Relapsed or Refractory Wilms' Tumor or Clear Cell Sarcoma of the Kidney
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CCLG-UKWR; CDR0000068913 (Registry Identifier: PDQ (Physician Data Query)); EU-20127
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2009-06

CONDITIONS: Kidney Cancer
Keywords: recurrent Wilms tumor and other childhood kidney tumors; clear cell sarcoma of the kidney
MeSH Terms: conditions — Kidney Neoplasms; Wilms Tumor | interventions — Dactinomycin; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Melphalan; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: dactinomycin
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: melphalan
Drug: vincristine sulfate
Procedure: autologous bone marrow transplantation
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: This phase II trial is studying how well chemotherapy followed by surgery and radiation therapy with or without stem cell transplant work in treating patients with relapsed or refractory Wilms' tumor or clear cell sarcoma of the kidney.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine survival rates of patients with relapsed or refractory Wilms' tumor or clear cell sarcoma of the kidney treated with chemotherapy followed by surgical resection and adjuvant radiotherapy with or without autologous stem cell rescue.
* Determine the efficacy and toxicity of these regimens in these patients.
* Determine prognostic variables in patients treated with these regimens.

OUTLINE: Patients are assigned to one of three treatment regimens.

* Regimen A (patients with initial stage I tumors previously treated with vincristine with or without dactinomycin with relapse at least 6 months after diagnosis): Patients receive vincristine IV once weekly on weeks 1-10 and then every 3 weeks during weeks 11-52, dactinomycin IV every 3 weeks during weeks 1-52, and doxorubicin IV over 6 hours every 3 weeks during weeks 1-34 (weeks 1-28 if pulmonary radiotherapy is planned). Patients undergo surgical resection and radiotherapy after 6 weeks of therapy.
* Regimen B (patients with initial stage II tumors previously treated with vincristine and dactinomycin with relapse at least 6 months after diagnosis): Patients receive cyclophosphamide IV twice daily on days 1-2 and 22-23, etoposide IV over 1 hour on days 1-3, and doxorubicin IV over 6 hours on days 22 and 23. Treatment repeats every 42 days for a total of 4 courses. Patients undergo surgical resection and radiotherapy after 2 courses of chemotherapy. Patients not achieving complete response after 4 courses of chemotherapy undergo autologous bone marrow transplantation as in regimen C.
* Regimen C (all other patients in first relapses OR with progression on first-line therapy OR in second or subsequent relapse previously treated on regimens A and B): Patients receive carboplatin IV over 1 hour on day 1, etoposide IV over 2 hours on days 1-3 and 22-24, and cyclophosphamide IV twice daily on days 22 and 23. Treatment repeats every 42 days for a total of 3 courses. Patients may undergo surgical resection prior to stem cell rescue. Beginning within 6 weeks after completion of chemotherapy, patients receive melphalan IV on day -1. Autologous peripheral blood stem cells or bone marrow is reinfused on day 0. Patients undergo radiotherapy after transplantation.

Patients are followed every 8 weeks for 1 year, every 12 weeks for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 75 patients (25 for regimens A and B and 50 for regimen C) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Wilms' tumor or clear cell sarcoma of the kidney, meeting 1 of the following criteria:

  * First relapse
  * Refractory (progression during first-line therapy)
* Patients in second and subsequent relapses allowed if previously treated with vincristine, dactinomycin, and doxorubicin combination chemotherapy (VCR/DACT/DOX)
* Metachronous tumors in the contralateral kidney allowed if previously treated with VCR/DACT/DOX
* No rhabdoid tumor of the kidney
* Previously treated on UK Wilms' tumor study

PATIENT CHARACTERISTICS:

Age:

* Under 18

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* See Disease Characteristics

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2001-05; Primary Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Unified treatment strategy
Improvement of current survival rates
Efficacy and toxicity
Prognostic variables

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Hale, MD, Study Chair — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - University College of London Hospitals, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland